CLINICAL TRIAL: NCT03933098
Title: A Phase III Multicenter, Observer-Blinded, Randomized, Active Controlled, Immune Non-inferiority and Safety Study of Vi-DT Vaccine Compared to Typbar TCV® in Healthy 6 Months-45 Years Aged Nepalese Participants.
Brief Title: Immune Non-inferiority and Safety of a Vi-DT Typhoid Conjugate Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI T003
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Typhoid
Keywords: Typhoid conjugate vaccine; Vi-DT; Safety; Immunogenicity
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Participants age 6 months to 45 years
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is observer blind:
  1. Vaccine administrator and vaccine safety evaluator at site will be two distinct persons.
  2. Laboratory personnel who analyzes immunogenicity at sponsor is also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test group A: Lot 1 Vi-DT (typhoid conjugate vaccine) (Experimental): One dose of Vi-DT (typhoid conjugate vaccine) Lot 1 will be administrated intramuscularly at Enrollment visit (Day 0).
  MR for age group at 9-15 months.
  Interventions: Biological: Test Vaccine Vi-DT Typhoid conjugate
- Test group B: Lot 2 Vi-DT (typhoid conjugate vaccine) (Experimental): One dose of Vi-DT (typhoid conjugate vaccine) Lot 2 will be administrated intramuscularly at Enrollment visit (Day 0).
  MR for age group at 9-15 months.
  Interventions: Biological: Test Vaccine Vi-DT Typhoid conjugate
- Test group C: Lot 3 Vi-DT (typhoid conjugate vaccine) (Experimental): One dose of Vi-DT (typhoid conjugate vaccine) Lot 3 will be administrated intramuscularly at Enrollment visit (Day 0).
  MR for age group at 9-15 months.
  Interventions: Biological: Test Vaccine Vi-DT Typhoid conjugate
- Test group D: Typbar TCV (Active Comparator): One dose of Typbar TCV will be administrated intramuscularly at Enrollment visit (Day 0).
  MR for age group at 9-15 months.
  Interventions: Biological: Control Vaccine Typbar TCV®

INTERVENTIONS:
Biological: Test Vaccine Vi-DT Typhoid conjugate — * Manufacturer: SK Bioscience Co., Ltd.
  * Ingredient: Purified Vi-polysaccharide conjugated to diphtheria toxoid
  * Dose: 25 µg of Vi polysaccharide/0.5 mL, presented in 3 mL multi-dose glass vial
  Other Names: Vi-DT Typhoid conjugate vaccine
  Arms: Test group A: Lot 1 Vi-DT (typhoid conjugate vaccine); Test group B: Lot 2 Vi-DT (typhoid conjugate vaccine); Test group C: Lot 3 Vi-DT (typhoid conjugate vaccine)
Biological: Control Vaccine Typbar TCV® — * Manufacturer: Bharat Biotech
  * Ingredient: Purified Vi capsular polysaccharide of Salmonella Ty2 conjugated to tetanus toxoid protein
  * Dose: 0.5 ml
  Other Names: Typbar TCV®
  Arms: Test group D: Typbar TCV

SUMMARY:
This is a Multicenter, observer-blinded, randomized, Active controlled, Phase 3 study in healthy 6 months to 45 years aged Nepalese at the time of the first vaccine dose.

The study objectives are:

I. Demonstrate non-inferiority of Vi-DT compared to Typbar TCV® as measured by seroconversion rates of anti-Vi IgG ELISA antibody titers, 4 weeks after single dose (pooled immunogenicity of three lots of Vi-DT)

II. Demonstrate the equivalence of immunogenicity as measured by anti-Vi IgG GMT of three lots of Vi-DT vaccine 4 weeks after single dose.

DETAILED DESCRIPTION:
Subjects will be stratified according to age. The study procedure is as follows:

Visit 1 (day-1 to -7): Screen participants by medical/medications history, physical examination, Vital signs, Urine pregnancy test (UPT)

Visit 2 (day 0): Enroll, randomize and administer vaccine to eligible participants and assess participant safety by physical examination and Vital signs, Collect blood for immunogenicity assessments.

Visit 3 (day 7): Check solicited adverse reaction 7 days post vaccination and Assess participant safety by physical examination and Vital signs

Visit 4 (day 28): Assess participant safety by physical examination and Vital signs, Collect blood for immunogenicity assessments

Visit 5 (day 84): Assess participant safety by physical examination and Vital signs

Visit 6 (day 168): Assess participant safety by physical examination and Vital signs, Collect blood for immunogenicity assessments, and fill in study completion form in the absence of any safety concern.

This study is observer-blind: vaccine administrator and vaccine safety evaluator will be two distinct persons to avoid bias of safety assessment. Trial staff other than the vaccine administrator.

For retention: After vaccination, field health worker/designee will contact participant every day till Day 7 by physical visit or by phone call. Follow-up reminder calls will be done very frequently as per discretion of study staff until 24 weeks for all participant to assess participant safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants 6 months to 45 years of age at enrollment
2. Participants/Parents/LAR who have voluntarily given informed consent/assent
3. Participants/Parents/LAR willing to follow the study procedures of the study and available for the entire duration of the study

Exclusion Criteria:

1. Child with a congenital abnormality
2. Subject concomitantly enrolled or scheduled to be enrolled in another trial
3. Known history of immune function disorders including immunodeficiency diseases (Known HIV infection or other immune function disorders)
4. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs
5. Receipt of blood or blood-derived products in the past 3 months
6. Subject with a previously ascertained or suspected disease caused by S. Typhi
7. Subject who have had household contact with/and or intimate exposure to an individual with laboratory-confirmed S. Typhi
8. Individual who has previously received a typhoid vaccine
9. Subject who has received or is expected to receive other vaccines from 1 month prior to IP vaccination to Visit 4 (approx.1 month post IP) except PVC booster as per EPI schedule
10. Known history or allergy to vaccines or other medications
11. History of uncontrolled coagulopathy or blood disorders
12. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the subject and interfere with the assessment of the study objectives
13. Any female participant who is lactating, pregnant* or planning for pregnancy during the course of study period
14. Participants/Parents/LAR planning to move from the study area before the end of study period
15. As per Investigator's medical judgement individuals could be excluded from the study inspite of meeting all inclusion/exclusion criteria mentioned above

    Temporary Contraindication
16. Acute illness, in particular infectious disease or fever (axillary temperature ≥37.5°C), within three days prior to enrolment and vaccination.

    * Urine pregnancy test (UPT) will be performed in all married females prior to injection

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate1 | 4 weeks (28 days) after vaccination of Vi-DT(pooled)/ Typbar TCV® compared to baseline (D0)
  Defined as a 4-fold increase of serum anti-Vi IgG antibody titer
Geometric Mean Titers (GMT)1 | 4 weeks after vaccination of Vi-DT
  Measurement of the Geometric Mean Titers (GMT) following 4 weeks after vaccination of three lots of Vi-DT

SECONDARY OUTCOMES:
Geometric Mean Titers (GMT) 2 | 4 weeks and 24 weeks after vaccination of Vi-DT(pooled)/ Typbar TCV®
  Measurement of the Geometric Mean Titers (GMT) following 4 weeks (28 days) and 24 weeks(168 days) after vaccination of Vi-DT (pooled)/ Typbar TCV®
Seroconversion rate 2 | 24 weeks (168 days) after vaccination of Vi-DT(pooled)/ Typbar TCV® compared to baseline (D0).
  Defined as a 4-fold increase of serum anti-Vi IgG antibody titer
Seroconversion rate 3 | 4 weeks (28 days) after vaccination of Vi-DT(pooled)
  Definded as a Seroconversion rates of anti-Vi IgG ELISA antibody titers after vaccination of three lots of Vi-DT.
Seroconversion rate 4 | 4 weeks (28 days) after vaccination of Vi-DT(pooled)
  Definded as a Seroconversion rates of anti-Vi IgG ELISA antibody titers at 4 weeks (28 days) after vaccination of three lots of Vi-DT in each age strata
Seroconversion rate 5 | 4 weeks (28 days) after vaccination of MR compared to baseline (D0)
  Definded as IgG ELISA antibody titers for Measles (M), and Rubella (R) following single dose of MR a vaccine at baseline D0 and 4 weeks
Safety endpoints for solicited adverse events (reactogenicity) | 7days after vaccination of Vi-DT(pooled)/ Typbar TCV®
  Proportion of participants with local and systemic solicited adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Kumar Rai, MD, Principal Investigator — Kanti Children's Hospital
Locations (4):
- Nepal (4):
  - Nepalgunj medical college, Bānke, City- Nepalgunj
  - B.P.Koirala Institute of Health Sciences, Rautahat, Dharan
  - Dhulikhel Hospital, Kavre, Dhulikhel
  - Kanti Children's Hospital, Kathmandu, Sukedhara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar Rai G, Saluja T, Chaudhary S, Tamrakar D, Kanodia P, Giri BR, Shrestha R, Uranw S, Kim DR, Yang JS, Park IY, Kyung SE, Vemula S, Reddy E J, Kim B, Gupta BP, Jo SK, Ryu JH, Park HK, Shin JH, Lee Y, Kim H, Kim JH, Mojares ZR, Wartel TA, Sahastrabuddhe S. Safety and immunogenicity of the Vi-DT typhoid conjugate vaccine in healthy volunteers in Nepal: an observer-blind, active-controlled, randomised, non-inferiority, phase 3 trial. Lancet Infect Dis. 2022 Apr;22(4):529-540. doi: 10.1016/S1473-3099(21)00455-2. Epub 2021 Dec 20. PMID 34942090